CLINICAL TRIAL: NCT02407964
Title: A Retrospective Epidemiologic Study on Incidence and Treatment Status of Hospitalized Drug Induced Liver Injury Patients in Mainland China
Brief Title: A Retrospective Study on Drug Induced Liver Injury in China
Acronym: DILI-R
Status: Completed | Type: Observational
Sponsor: Drug Induced Liver Disease Study Group (Other)
Collaborators: Unimed Scientific Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012ZX09303-001
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Drug-Induced Liver Injury
Keywords: Drug-Induced Liver Injury; DILI
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center, open-enrollment, retrospective, non-interventional epidemiologic study without any clinical treatment. Its primary objective is to understand 1) incidence of drug-induced liver injury, including incidences among all the hospitalized patient, among patients in department of hepatic diseases, digestive diseases, oncology, hematology etc., individually; 2) epidemiologic characteristics of drug-induced liver injury, including suspected medications, clinical types, histological characteristics, severity and outcomes.

DETAILED DESCRIPTION:
This is a multi-center, open-enrollment, retrospective, non-interventional epidemiologic study without any clinical treatment. Its primary objective is to understand 1) incidence of drug-induced liver injury, including incidences among all the hospitalized patient, among patients in department of hepatic diseases, digestive diseases, oncology, hematology etc., individually; 2) epidemiologic characteristics of drug-induced liver injury, including suspected medications, clinical types, histological characteristics, severity and outcomes.

It investigates medical records of patients who were hospitalized during 2012 to 2014. Those patients should be diagnosed as drug-induced liver injury, drug-induced liver disease, drug-induced hepatitis, drug-induced hepatocirrhosis, drug-induced hepatic failure, or any other similar diagnosis of drug-induced liver injury nature.

ELIGIBILITY:
Inclusion Criteria:

* Any hospitalized patients who were diagnosed as drug-induced liver injury, drug-induced liver disease, drug-induced hepatitis, drug-induced hepatocirrhosis, drug-induced hepatic failure, or any other similar diagnosis of drug-induced liver injury nature.
* The drug-induced liver injury and similar diagnosis were not excluded the possibility of drug-induced nature.

Exclusion Criteria:

* Confirmed non-drug induced liver injury.
* Insufficient clinical data supporting the diagnosis of drug-induced liver injury.
* Liver injury resulted from poisons and chemicals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were hospitalized during 2012 to 2014.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
diagnosis of drug-induced liver injury | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Mao, MD, Study Chair — RenJi Hospital; Chengwei Chen, MD, Study Chair — No. 85 Hospital of PLA
Locations (371):
- China (371):
  - Department of gastroenterology,the second hospital of Shanxi medical university, Taiyuan, Shanxi
  - Department of gastroentrology of Ankang city central hospital, Ankang
  - Department of gastroenterology of Anqing municipal hospital, Anqing
  - Department of infectious disease of Anqing municipal hospital, Anqing
  - Department of tuberculosis of Baoding infectious disease hospital, Baoding
  - Department of gastroentrology,the third hospital of PLA, Baoji
  - Department of infectious disease of Baoji No.2 people's hospital, Baoji
  - Department of infectious disease,the third hospital of PLA, Baoji
  - Department of tuberculosis,the third hospital of PLA, Baoji
  - Department of lymph&breast of Baotou tumor hospital, Baotou
  - Department of breast disease,Tongzhou matermal&child health hospital of Beijing, Beijing
  - Department of gastroenterology of Beijing Huairou hospital, Beijing
  - Department of Hepatology of Beijing Ditan Hospital Capital Medical University, Beijing
  - Department of hepatology of Peking university people's hospital, Beijing
  - Department of infection of Peking university first hospital, Beijing
  - Non infedtious liver disease diagnosis and treatment center,302 military hospital of China, Beijing
  - Department of gastroenterology,the first affiliated hospital of Bengbu medical college, Bengbu
  - Department of infectious disease,the first affiliated hospital of Bengbu medical college, Bengbu
  - Department of infectious disease,the No.123 hospital of PLA, Bengbu
  - Department of gastroenterology of Cangzhou central hospital, Cangzhou
  - Department of gastroenterology,the fourth hospital of Jilin university, Changchun
  - Department of infectious disaese,the fourth hospital of Jilin unversity, Changchun
  - Department of infectious disease of Changchun infectious disease hospital, Changchun
  - Department of rhenmatism,the affiliated hospital to Changchun University of Chinese medicine, Changchun
  - Department of infectious disease,people's hospital Changji hui autonomous prefecture Xinjiang, Changji
  - 2st department of hepatology,the first hospital of Changsha, Changsha
  - 5st internal meidcine of Hunan chest hospital, Changsha
  - Department of breast disease,the affiliated cancer hospital of Xiangya school, Changsha
  - Department of infectious disease of Hunan provincial people's hospital, Changsha
  - Department of infectious disease of Xiangya hospital central south university, Changsha
  - Department of infectious disease,the second Xiangya hospital of central south university, Changsha
  - Department of infectious disease,the third Xiangya hospital of central south university, Changsha
  - Department of tuberculosis of Changsha central hospital, Changsha
  - Department of infectious disease,Heping hospital affiliated to Changzhi medical university, Changzhi
  - Department of hepatology of Chengdu tenth people's hospital, Chendu
  - Department of gastroenterlogy,affiliated hospital of Chenfdu University, Chengdu
  - Department of gastroenterology,the 416th hospital of CNNC, Chengdu
  - Department of gastroenterology of Chenzhou No.1 people's hospital, Chenzhou
  - Department of hepatology of Chenzhou No.2 people's hospital, Chenzhou
  - Department of infectious disease,the fourth people's hospital of Chenzhou, Chenzhou
  - Department of infectious disease,the people's hospital of Chizhou, Chizhou
  - Department of hepatology,Chongqing hospital of TCM, Chongqing
  - Department of infectious disease of southwest hospital, Chongqing
  - Department of infectious disease,the second affiliated hospital of Chongqing medical university, Chongqing
  - Department of gastroenterology of Daqing oilfield general hospital, Daqing
  - Department of infectious disease of Daqing second hospital, Daqing
  - Department of hepatology of Datong fourth people's hospital, Datong
  - Department of gastroenterology,Qilu hospital of Shandong university, Dongying
  - Department of infectious disease of Shengli oilfield general hospital, Dongying
  - Department of infectious disease ，Shengli hospital of Shengli oilfield administration, Dongying
  - Department of infectious disease of Shanxi province Fenyang hospital, Fenyang
  - Department of infectious disease of Foshan first people's hospital, Foshan
  - Department of infectious disease of Fujian province Fuqing city hospital, Fuqing
  - Department of hepatologym,No.2 people's hospital of Fuyang, Fuyang
  - Department of hepatic-biliary medicine,Fuzhou general hospital of Nanjing military command, Fuzhou
  - Department of hepatic-biliary medicine,No.476 hospital of PLA, Fuzhou
  - Department of hepatology of Fuzhou infectious disease hospital, Fuzhou
  - Department of digestive of Guangdong general hospital, Guangdong
  - Deaprtment of gastroenterology of Guangzhou first people's hospital, Guangzhou
  - Department of gastroenterology of Guagdong general hospital, Guangzhou
  - Department of gsatroenterology of Sun Yat-sen memorial hspital, Sun Yat-sen university, Guangzhou
  - Department of infectious disease of Guangzhou women&children medical center, Guangzhou
  - Department of infectious disease,Nanfang hospital of southern medical university, Guangzhou
  - Department of science education&information of Guangzhou Huiai hospital, Guangzhou
  - Department of hematology,the affiliated hospital of Guiyang medical university, Guiyang
  - Department of infectious disease of Guizhou provincial people's hospital, Guiyang
  - Department of infectious disease,the affiliated hospital of Guiyang medical university, Guiyang
  - 10st department of internal medicine of Heilongjiang province center for tuberculosis control and prevention, Haerbin
  - 1st mepartment of internal medicine Heilongjiang province center for tuberculosis control and prevention, Haerbin
  - 4st department of internal medicine of Heilongjiang province center for tuberculosis control and prevention, Haerbin
  - 5st department of internal medicine of Heilongjiang province center for tuberculosis control and prevention, Haerbin
  - 7st department of internal medicine of Heilongjiang province center for tuberculosis control and prevention, Haerbin
  - 8st department of internal medicine of Heilongjiang province center for tuberculosis control and prevention, Haerbin
  - 9st department of internal medicine of Heilongjiang province center for tuberculosis control and prevention, Haerbin
  - Department of infectious disease,No.211 hospital of PLA, Haerbin
  - Department of infectious disease,the first affiliated hosptal of Haerbin medical university, Haerbin
  - Department of infection of Hainan general hospital, Hainan
  - Department of infectious disease of Hangzhou Xiaoshan district first people's hospital, Hangzhou
  - Department of infectious disease of Sir Run Run Shaw hospital,Zhejiang unicersity school of medicine, Hangzhou
  - 1st department of respiration of Hanzhong second people's hospital, Hanzhong
  - Department of infection of Hanzhou first people's hospital, Hanzhou
  - Department of gastroenterology,the first affiliated hospital of Anhui medical university, Hefei
  - Department of infectious disease of Anhui provincial hospital, Hefei
  - Department of infectious disease of Hefei infectious disease hospital, Hefei
  - Department of infectious disease,No.105 hospital of PLA, Hefei
  - Department of infectious disease,the first affiliated hospital of Anhui university of Chinese medicine, Hefei
  - Department of hematology of First affiliated hospital,Heilongjiang university of Chinese medicine, Heilongjiang
  - Department of infectious disease,the first affiliated hospital of university of south China, Hengyang
  - Department of hepatology of Hohhot second hospital, Hohhot
  - Department of hepatology of Huai'an No.4 people's hospital, Huai'an
  - department of oncology,Huaiyin hospital of Huai'an city, Huai'an
  - Department of infectious disease of Yili friendship hospital, Huiyuan
  - Department of infectious disease,people's hospital of Puluo county, Huizhou
  - Department of oncology,people's hospital of Puluo county, Huizhou
  - Department of gastroenterology of inner mongolia forestry general hospital, Inner Mongolia
  - Department of hepatology of Inner Mongolia international Mongolian medicine hospital, Inner Mongolia
  - Department of hepatology of No.253 hospital of the PLA, Inner Mongolia
  - Department of infection, the affiliated hospital of inner mongolia medical hospital, Inner Mongolia
  - Department of infection,the first affiliated hospital of Baotou medical university, Inner Mongolia
  - Department of infectious disease of inner mongolia people's hospital, Inner Mongolia
  - Department of tuberculosis of The Inner Mongolia Autonomous Region fourth hospital, Inner Mongolia
  - Department of hematology, first affiliated hospital of Jiamusi university, Jiamusi
  - Internal medicine,the 404 hospital of China national nuclear, Jiayuguan
  - Department of gastroenterology of Beihua university affiliated hospital, Jilin
  - Department of gastroenterology,hepatology hospital of Jilin province, Jilin
  - Department of gastroentrology of Jilin integrated TCM&western medicine hospital, Jilin
  - Department of hepatology,hepatology hospital of Jilin province, Jilin
  - Department of hepatology,the first hospital oof Jilin university, Jilin
  - Department of infectious disease of Beihua university affiliated hospital, Jilin
  - 1st department of hepatology of Jinan hospital for infectious disease, Jinan
  - Department of endocrinology of Shangdong provincial hospital, Jinan
  - Department of gastroenterology of Jinan central hospital, Jinan
  - Department of gastroenterology,Qilu hospital of Shandong university, Jinan
  - Department of gastroenterology,the second hospital of Shandong university, Jinan
  - Department of hepatology of Shandong province Qianfoshan hospital, Jinan
  - Department of hepatology of Shandong provincial hospital of Chinese medicine, Jinan
  - Department of rheumatology of Shandong provincial hospital, Jinan
  - Internal medicine of Jinan city Lixia district people's hospital, Jinan
  - Department of infectious disease of Jincheng anthracite mining group general hospital, Jincheng
  - Department of infectious disease of Zezhou county people's hospital, Jincheng
  - 2st department of hepatology of Jingmen No.2 people's hospital, Jingmen
  - Department of gastroenterology of Jingmen No.1 people's hospital, Jingmen
  - Department of gastroenterology ward 2 of Jingmen No.1 people's hospital, Jingmen
  - Department of infectious disease of Jingmen No.2 people's hospital, Jingmen
  - 1st internal medicine of Jingzhou hospital for infectious disease, Jingzhou
  - Department of infectious disease of Jingzhou central hospital, Jingzhou
  - Department of gastroenterology of Jinzhong City Yuci district people's hospital, Jinzhong
  - Department of gastroenterology of Qixian county people's hospital, Jinzhong
  - Department of gastroenterology,the second people's hospital of Jinzhong, Jinzhong
  - Department of gastroentrology,the first people's hospital of Jinzhong, Jinzhong
  - Department of infectious disease,the first affiliated hospital of Henan university, Kaifeng
  - Department of infectious disease of Kashgar prefecture first people's hospital, Kashgar
  - Department of gastroenterology of Xishan district people's hospital, Kunming
  - Department of gastroenterology of Yunnan first people's hospital, Kunming
  - Department of gastroenterology,the first affiliated hospital of Kunming medical university, Kunming
  - Department of gastroentrology,the first hospital of Kunming, Kunming
  - Department of infectious disease,Kunming general hospital of Chengdu military, Kunming
  - Department of infectious disease,the first affiliated hospital of Kunming medical university, Kunming
  - Department of rheumatology of Yunnan first people's hospital, Kunming
  - Hepatology center,the second affiliated hospital of Kunming medical university, Kunming
  - Department of hepatology, Gansu provincial hospital of TCM, Lanzhou
  - Department of infectious disease of Lanzhou military general hospital, Lanzhou
  - Department of infestious disease,the first hospital of Lanzhou university, Lanzhou
  - outpatient of pulmonary hospital of Lanzhou, Lanzhou
  - Department of infectious disease of Leqing people's hospital, Leqing
  - Department of hepatology of Liaocheng city infectious disease hospital, Liaocheng
  - Department of hepatology &respiration of Linfen infectious disease hospital, Linfen
  - Department of endocrinolnogy of Linyi people's hospital, Linyi
  - Department of hepatology of Linyi people's hospital, Linyi
  - Department of tuberculosis of Linyi people's hospital, Linyi
  - Department of gastroenterology of Lu'an people's hospital, Lu'an
  - Department of gastroenterology of Luoyang third people's hospital, Luoyang
  - Department of infectious disease of Luoyang central hospital, Luoyang
  - Department of infectios disease,the affiliated hospital of southwest hospital, Luzhou
  - Department of hepatology ward 1 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of hepatology ward 2 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of hepatology wardf 10 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of hepatology wardf 3 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of hepatology wardf 4 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of hepatology wardf 9 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of tuberculosis of ward 11 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of tuberculosis ward 5 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of tuberculosis ward 6 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of tuberculosis ward 7 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of tuberculosis ward 8 of Mudanjiang Kangan hospital, Mudanjiang
  - Department of gastroenterology of Jiangxi provincial people's hospital, Nanchang
  - Department of gastroenterology of the second affiliated hospital to Nanchang university, Nanchang
  - Department of tuberculosis of Jiangxi provincial chest hospital, Nanchang
  - Deparment of oncology, Nanjing hospital of TCM, Nanjing
  - Department of hematology of Nanjing Jiangning hospital, Nanjing
  - Department of hematology, Jiangsu province hospital of TCM, Nanjing
  - Department of hepatology,No.81 hospital of PLA, Nanjing
  - Department of infection of Jiangsu province hospital, Nanjing
  - Department of infection of Nanjing drum tower hospital, Nanjing
  - Department of infection,the second hospital of Nanjing, Nanjing
  - Department of infectious disease of Nanjing Jiangbei people's hospital, Nanjing
  - Department of infectious,Jiangsu procince hospital of TCM, Nanjing
  - Department of oncology , Jiangning hospital of Nanjing city, Nanjing
  - Department on tuberculosis of Nanjing chest hospital, Nanjing
  - Department of gastroenterology,the first affiliated hospital of Guangxi medical university, Nanning
  - Department of hepatology,the first affiliated hospital of Guangxi university of Chinese medicine, Nanning
  - Department of oncology，the first affiliated hospital of Guangxi university of Chinese medicine, Nanning
  - Department of gastroenterology of Ningbo medical treatment center Lihuili hospital, Ningbo
  - Department of gastroenterology,Yinzhou hospital affiliated to medical school of Ningbo university, Ningbo
  - Department of hematology of Ningbo medical treatment center Lihuili hospital, Ningbo
  - Department of hepatology of Ningbo No.2 hospital, Ningbo
  - Department of hepatology,No.113 hospital of PLA, Ningbo
  - Department of psychiatry of Ningbo Kangning hospital, Ningbo
  - Department of infectious disaese of Erdos second people's hospital, Ordos
  - Department of oncology of Jungar Banner central hospital, Ordos
  - Department of tuberculosis of Pingdingshan third people's hospital, Pingdingshan
  - Department of gastroenterology of Jiangxi Pingxiang people's hospital, Pingxiang
  - Department of gastroenterology,Pingxiang city hospital of Chinese medicine, Pingxiang
  - Department of infedtious disease of Pingyang county hospital of Chinese medicine, Pingyang
  - Department of infectious disease,Puyang oilfield general hospital, Pujiang
  - Department of tuberculosis,the fifth people hospital of Puyang, Pujiang
  - Department of digestive,the affiliated hospital of Qingdao university, Qingdao
  - Department of endocrinology,the affiliated hospital of Qingdao university, Qingdao
  - Department of gastroenterology of Qingdao municipal hospital, Qingdao
  - Department of hepatology,the affiliated hospital of Qingdao university, Qingdao
  - Department of digestive of Qinghai provincial people's hospital, Qinghai
  - Department of hepatology,Qinghai province hospital for infectious disease, Qinghai
  - Deqpartment of gastroenterology of Qinghai university affiliated hospital, Qinghai
  - Department of gastroenterology,the third hosital of Qinhuangdao, Qinhuangdao
  - Department of hepatology,the third hospital of Qinhuangdao, Qinhuangdao
  - Department of infectious disease of Qiqihar infectious disease hospital, Qiqihar
  - Department og gastroenterology,the first hospital of Qiqihar city, Qiqihar
  - Department of infectious disease of Ruian people's hospital, Ruian
  - Department of gastroenterology of Sanmenxia central hospital, Sanmenxia
  - Department of hematology of Sanmenxia central hospital, Sanmenxia
  - Department of infectious disease of Sanmenxia central hospital, Sanmenxia
  - Department of gastroenterology,No.301 hospital Sanya branch, Sanya
  - Clinical research center for tuberculosis of Shanghai pulmonary hospital, Shanghai
  - Department of Digestive Diseases of Shanghai Tongji Hospital, Shanghai
  - Department of Digestive Diseases of The Renji Hospital, Shanghai
  - Department of digestive of Shanghai Tongji hospital, Shanghai
  - Department of gastroenterolgy of Huadong hispital affiliated to Fudan university, Shanghai
  - Department of gastroenterology,the affiliated Zhongshan hospital of Fudan university, Shanghai
  - Department of hepatocirrhosis of Shuguang hospital affiliated Shanghai University of T.C.M, Shanghai
  - Department of hepatology of No.85 hospital of PLA, Shanghai
  - Department of infection of No.85 hospital of PLA, Shanghai
  - Department of Infection of Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Department of infectious disease of Longhua hospital affiliated to Shianghai univesity of Chinese medicine, Shanghai
  - Department of infectious disease of Shanghai Songjiang district people's hospital, Shanghai
  - Department of infectious disease of Tongren hospital, Shanghai
  - Department of infectious disease,Huashan hospital affiliated to Fudan university, Shanghai
  - Department of oncology of Shanghai Putuo district central hospital, Shanghai
  - Department of oncology of the sixth people's hospital affiliated to Shanghai Jiaotong university, Shanghai
  - Department of pediatrics of Shanghai first people's hospital Songjiang branch, Shanghai
  - Department of digestive of the second affiliated hospital of Xi'an jiaotong university, Shangxi
  - Department of infection of the second affiliated hospital of Xi'an jiaotong university, Shangxi
  - Department of gastroenterology of Shanluo central hospital, Shanluo
  - Department of infectious disease of Shanluo central hospital, Shanluo
  - Department of infectious disease of Shaoxing central hospital, Shaoxing
  - Department of infectious disease of Shaoyang central hospital, Shaoyang
  - Department of infectious disease,Shengjing hospital of China medical university, Shenyang
  - Department of hepatology of Shenzhen third people's hospital, Shenzhen
  - Department of infectious disease of Shenzhen third people's hospital, Shenzhen
  - Department of pulmonary dedicine of Shenzhen third people's hospital, Shenzhen
  - Department of gastroenterology of Hebei general hospital, Shijiazhuang
  - Department of gastroenterology,the first hospital of Hebei medical university, Shijiazhuang
  - Department of hematology,the first hospital of Hebei medical university, Shijiazhuang
  - Department of hepatology,the first hospital of Hebei medical university, Shijiazhuang
  - Department of hepatology，the third hodpital of Hebei medical university, Shijiazhuang
  - Department of tuberculosis of Hubei province chest hospital, Shijiazhuang
  - 2st department of gastroenterology of Shiyan people's hospital, Shiyan
  - Department of infectious disease of Dongfeng company general hospital, Shiyan
  - Department of infectious disease of Taihe hospital, Shiyan
  - Department of tuberculosis of Xiyuan hospital of Shiyan city, Shiyan
  - Department of infestious disease,the first people's hospital of Shunde, Shunde
  - Department of gastroenterology of Songyuan central hospital, Songyuan
  - Department of hepatology of Jilin oilfiled general hospital, Songyuan
  - Department of infectious disease of Suzhou municipal hospital, Suzhou
  - Department of infectious disease,the fifth people's hospital of Suzhou, Suzhou
  - Department of i fectious disease of Taian city central hospital, Taian
  - Department of tuberculosis of Taian cancer hospital, Taian
  - 1st department of tuberculosis of Taiyuan fourth people's hospital, Taiyuan
  - Department of hepatology,Shanxi provincial hospital of Chinese medicine, Taiyuan
  - Department of tuberculosis of Taiyuan fourth people's hospital, Taiyuan
  - Department of hematology&oncology,Taizhou hospital of Zhejiang province, Taizhou
  - Department of infectious disease of Tianchang people's hospital, Tianchang
  - Department of hepatology of Tianjin first hospital, Tianjin
  - Department of hepatology of Tianjin third central hospital, Tianjin
  - Department of hepatology,first teaching hospital of Tianjin university, Tianjin
  - Department of hepatology,The affiliated hospital of logistics university of people's armed police force, Tianjin
  - Department of oncology of Tianjin medical university general hospital, Tianjin
  - Department of rheumatology of Tianjin first center hospital, Tianjin
  - Department of infestious disaese of Tibet autonomous prefecture people's hospital, Tibet
  - 1st department of oncology of Tonghua central hospital, Tonghua
  - 3st department of oncology of Tonghua central hospital, Tonghua
  - Department of oncology of Tonghua second people's hospital, Tonghua
  - Department of oncology&hematology of Tonghua people's hospital, Tonghua
  - Department of infectious disease of Tongliao infectious disease hospital, Tongliao
  - Department of hepatology of The Xinjiang production and construction Corps hospital, Ürümqi
  - Department of infectious disease of URUMQI friendship hospital, Ürümqi
  - 2st department of tuberculosis of Weifang No.2 people's hospital, Weifang
  - Department of gastroenterology of Weifang people's hospital, Weifang
  - Department of gastroenterology of Weihai central hospital, Weihai
  - Department of gastroenterology of Weihai municipal hospital, Weihai
  - Department of infectious disease of Weinan central hospital, Weinan
  - Department of infectious disease,the first people's hospital of Wenling, Wenling
  - Department of hematology of the first affiliated hospital of Wenzhou medical university, Wenzhou
  - Department of infectious disease of Wencheng county people's hospital, Wenzhou
  - Department of infectious disease,Wenshou hospital of Chinesemedicine, Wenzhou
  - Department of oncology of Wuhai people's hospital, Wuhai
  - 1st internal medicine of Wuhan institute for tuberculosis control, Wuhan
  - 3st internal medicine of Wuhan institute for tuberculosis control, Wuhan
  - 4st internal medicine of Wuhan institute for tuberculosis control, Wuhan
  - 5st internal medicine of Wuhan institute for tuberculosis control, Wuhan
  - Departmeent of gastroenterology of fifth hodpital in Wuhan, Wuhan
  - Department of gastroenterology of Wuhan integrated TCM&western medicine hospital, Wuhan
  - Department of gastroenterology of Wuhan union hospiital, Wuhan
  - Department of gastroenterology,the central hospital of Wuhan, Wuhan
  - Department of gastroenterology,Wuhan general hospital of Guangzhou military, Wuhan
  - Department of hepatology of Wuhan seventh hospital, Wuhan
  - Department of hepatology,Hubei provincial hospital of TCM, Wuhan
  - Department of hepatology,Wuhan general hospital of Guangzhou military, Wuhan
  - Department of infectious disease of Puren hospital, Wuhan
  - Department of infectious disease of Wuhan iron and steel(group) corp. staff hospital, Wuhan
  - Department of infectious disease of Wuhan iron and steel(group) Crop. second staff hospital, Wuhan
  - Department of infectious disease of Wuhan union hospital, Wuhan
  - Department of infectious disease(north fifth ward) of Wuhan medical treatment center, Wuhan
  - Department of infectious disease（north fourth ward） of Wuhan medical treatment center, Wuhan
  - Department of infectious disease（north sixth ward) of Wuhan medical treatment center, Wuhan
  - Department of infectious disease（south second ward） of Wuhan medical treatment center, Wuhan
  - Department of oncology,Renmin hospital of Hubei university, Wuhan
  - Department of tuberculosis(south fifth ward) of Wuhan medical treatment center, Wuhan
  - Department of tuberculosis(south first ward) of Wuhan medical treatment center, Wuhan
  - Department of tuberculosis(south fourth ward) of Wuhan medical treatment center, Wuhan
  - Department of tuberculosis(south sixth ward) of Wuhan medical treatment center, Wuhan
  - Department of gastroenterology,the first affiliated hospital of Wannan medical college, Wuhu
  - Department of oncology of Wuxi No.2 people's hospital, Wuxi
  - 1st internal medicine of Shangxi province tuberculosis prevention and treatment institute, Xi'an
  - 2st department of gastroenterology of Shaanxi provincial people's hospital, Xi'an
  - 3st internal medicine of Shanxi province tuberculosisi prevention and treatment institute, Xi'an
  - Department of gastroenterology of Xi'an children's hospital, Xi'an
  - Department of gastroenterology of Xijing hospital, Xi'an
  - Department of gastroenterology,No.451 hospital of PLA, Xi'an
  - Department of gastroenterology,the first affiliated hospital of Xi'an Jiaotong university, Xi'an
  - Department of infectious disease,the first affiliated hospital of Xiamen university, Xiamen
  - Departmenr of infectious disease,the first people's hospital of Xiangtan city, Xiangtan
  - Department of infectious disease of Xiangtan central hospital, Xiangtan
  - 2st department of gastroenterology of Xiangyang central hospital, Xiangyang
  - Department of gastroenterology B zone of Xiangyang No.1 people's hospital, Xiangyang
  - Department of gastroenterology of Xianyang central hosppital, Xianyang
  - Department of infectious disease of Xianyang central hospital, Xianyang
  - Department of infectious disease,the affiliated hospital of Shaanxi university of Chinese medicine, Xianyang
  - Department of tuberculosis of Xianyang central hospital, Xianyang
  - 2st department of oncology,Xinjiang Uyghur aotonomous region hospital of Chinese medicine, Xinjian
  - 1st department of oncology,Xinjiang Uyghur aotonomous region hospital of Chinese medicine, Xinjiang
  - 4st department of tuberculosis,chest hospital of Xinjiang Uyghur aotonomous region of the PRC, Xinjiang
  - Department of hepatology,Xinjiang Uyghur aotonomous region hospital of Chinese medicine, Xinjiang
  - Department of infectious disease of Xinjiang general hospital of CAPF, Xinjiang
  - Department of infectious disease of Xinjiang Uyghur aotonomous region people's hospital, Xinjiang
  - Department of infectious,the first affiliated hospital of Xinjiang medical university, Xinjiang
  - 2st department of infectious disease,the first affiliated hospital of Xinxiang medical university, Xinxiang
  - Department of gastroenterology,Xinyu hospital of Chinese medicine, Xinyu
  - Department of science education of Xinzhou city people hospital, Xinzhou
  - Department of infectious disease of Ya'an people's hospital, Ya'an
  - Department of gastroenterology of Yanan university affiliated hospital, Yanan
  - Department of respiration of Yanan university affiliated hospital, Yanan
  - Department of psychiatry of Yanbian brain hospital, Yanbian
  - Department of hepatology of Yancheng second people's hospital, Yancheng
  - Department of infectious disease of Yancheng city No.1 people's hospital, Yancheng
  - Department of gastroenterology of Yangguan coalmine group general hospital, Yangquan
  - Department of digestive of northern Jiangsu people's hospital, Yangzhou
  - Department of infectious disease,the third hospital of Yangzhou city, Yangzhou
  - Department of oncology of Northern Jiangsu peolple's hospital, Yangzhou
  - Department of gastroenterology of Yanji hospital, Yanji
  - Department of gastroenterology of Yichang first people's hospital, Yichang
  - Department of infectious disease of China Gezhouba group central hospital, Yichang
  - Department of infectious disease of Yichang central people's hospital, Yichang
  - Department of infectious,general hospital of Ningxia medical university, Yinchuan
  - Department of hepatology of Yiyang infectious disease hospital, Yiyang
  - Department of infectious disease,the first hospital of Yulin, Yulin
  - Department of hepatology of Yuncheng infectiuos disease hospital, Yuncheng
  - Department of infectious of Yuyao people's hospital, Yuyao
  - 1st department of respiration of Zhengzhou sixth people's hospital, Zhengzhou
  - 7st department of respiration of Zhengzhou sixth people's hospital, Zhengzhou
  - Department of digestive of Henan provincial people's hospital, Zhengzhou
  - Department of gastroenterology,the fifth affiliated hospital of Zhengzhou, Zhengzhou
  - Department of gastroenterology,the first affiliated hospital of Henan university of TCM, Zhengzhou
  - Department of gastroentrology of Zhengzhou central hospital, Zhengzhou
  - Department of hepatic-biliary meidicine,No.153 hospital of PLA, Zhengzhou
  - Department of infection,the first affiliated hospital of Zhengzhou university, Zhengzhou
  - Department of infectious disaese of Henan provincial people's hospital, Zhengzhou
  - Department of tuberculosis of Zhengzhou 6th people's hospital, Zhengzhou
  - lienic-gastric-hepatic medicine,Zhengzhou hospital of Chinese medicine, Zhengzhou
  - Department of infectious disease of Zhuzhou central hospital, Zhuzhou
  - Department of digestive of Yiyuan county people's hospital, Zibo
  - Department of rheumatology,central hospital of Zibo, Zibo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Zhang J, Xu X, Fang W, Qu S, Jin F, Zhou J, Han X, Raza HK, Li X, Mao Y. Hugan tablets for the treatment of RUCAM based drug-induced liver injury: a propensity score matching analysis using a nationwide database. Expert Rev Clin Pharmacol. 2021 Dec;14(12):1543-1550. doi: 10.1080/17512433.2021.1981859. Epub 2021 Sep 22. PMID 34521298